CLINICAL TRIAL: NCT00056251
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of RTX Topical Solution in Patients With Interstitial Cystitis
Brief Title: Interstitial Cystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JIC01
Record Dates: First submitted 2003-03-07; First posted 2003-03-10 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial Cystitis; Bladder
MeSH Terms: conditions — Cystitis, Interstitial | interventions — epicatechin gallate; Hematologic Tests; Cystoscopy

INTERVENTIONS:
Procedure: H&P; ECG; Blood tests; voiding diary; Cystoscopy

SUMMARY:
Patients with interstitial cystitis who meet eligibility requirements will be randomized to one of four treatment arms (3 RTX, Placebo). Study drug is administered as a single instillation within the urinary bladder. Study duration is 12 weeks.

DETAILED DESCRIPTION:
RATIONALE:

Topical resiniferatoxin (RTX) administrated to the bladder may be effective in decreasing the symptoms associated with interstitial cystitis through its action on pain sensing neurons.

PURPOSE:

Randomized, double-blind, placebo-controlled, Phase 2 trial to determine the safety and efficacy of RTX in patients with interstitial cystitis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Have IC that meets disease diagnostic criteria as defined by a history of the following:
* Cystoscopy/hydrodistension with a diagnosis of IC confirmed by findings of Hunner's ulcer or glomerulation
* Symptoms of bladder pain and urinary urgency for at least 6 months
* Urinary frequency while awake at least 8 times a day while awake
* Nocturia at least twice a night
* Symptoms not significantly relieved by antimicrobial agents, anticholinergic drugs, or antispasmodics
* Have IC that in the judgment of the investigator has been stable in the previous 30 days
* Have IC-related pain despite current therapy, defined as a score of 4 or greater [(on a scale from 0 (none) to 9 (severe)] on average over the past month and confirmed by the voiding diary collected at Visit 2
* Have at least one voided volume ≥ 75 cc in a 24 hour period, confirmed by the voiding diary collected at Visit 2
* Patients of childbearing potential must agree to use an acceptable form of contraception (oral contraceptives, intrauterine device or double barrier methods) from Visit 1 through Visit 6
* Provide signed informed consent

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Presence of ulcers on the pre-treatment cystoscopy
* Intravesical therapy or bladder hydrodistention within the previous 60 days
* Initiation of pentosan polysulfate sodium (Elmiron®) within the previous 16 weeks
* Use of fentanyl patches, morphine sulfate, methadone or B&O supprettes within the previous 30 days.
* Previous augmentation cystoplasty, cystectomy or cystolysis, neurectomy (i.e., hypogastric nerve plexus ablation) or implanted peripheral nerve stimulator which has affected bladder function
* History of ureteral reflux. Patients with a history of childhood urinary tract infections, recurrent urinary tract infections as an adult (defined as >3 culture documented episodes within the previous 12 months), or pyelonephritis at any time must have a cystourethogram to rule out ureteral reflux.
* Evidence of renal impairment (creatinine > 2 times the upper limit of normal at Visit 1), hepatic impairment (AST or ALT > 3 times the upper limit of normal at Visit 1), clinically significant cardiovascular, respiratory, or psychiatric diseases
* Any condition that in the judgment of the investigator would interfere with the patient's ability to provide informed consent, comply with study instructions, place the patient at increased risk, or which might confound the interpretation of the study results
* Treatment with a drug or medical device that has not received regulatory approval within the previous 30 days
* Investigators, study staff and their immediate families. Immediate family is defined as current spouse, parent, natural or legally adopted child (including a stepchild living in the investigator's household), grandparent, or grandchild.
* Previously completed or withdrawn from this study
* Urinary tract or prostatic infection within the past 3 months before study entry
* Active genital herpes or vaginitis
* Urethral diverticulum
* Uterine, cervical, vaginal, or urethral cancer within the past 5 years before study entry
* History of cyclophosphamide or chemical cystitis, urinary tuberculosis or radiation cystitis
* History of bladder tumors (benign or malignant)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-01; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Lyn Frumkin, M.D., Ph.D., Study Director — ICOS Corporation, (425) 415-5571, lfrumkin@icos.com
Locations (24):
- United States (24):
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Citrus Valley Medical Research, Inc., Glendora, California
  - Center for Urological Research, La Mesa, California
  - Atlantic Urological Medical Group, Long Beach, California
  - Stanford University Medical Center, Stanford, California
  - Colorado Gynecology & Continence Center, Denver, Colorado
  - dba Genitourinary Surgical Consultants, PC, Denver, Colorado
  - The Connecticut Clinical Research Center-Urology Specialist, Waterbury, Connecticut
  - Advanced Research Institute, New Port Richey, Florida
  - Georgia Urology, Atlanta, Georgia
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Urology of Indiana, LLC, Indianapolis, Indiana
  - KU Medical Center Research Institute, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - Michigan William Beaumont Hospital, Royal Oak, Michigan
  - St. Louis Urological Surgeons, St Louis, Missouri
  - Michael Kaplan, MD, Ltd., Henderson, Nevada
  - The Urology Center, Greensboro, North Carolina
  - Urologic Specialists of Oklahoma, Tulsa, Oklahoma
  - Oregon Urology Specialists, Eugene, Oregon
  - Pennsylvania Graduate Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology San Antonio, San Antonio, Texas
  - Integrity Medical Research, LLC, Seattle, Washington